CLINICAL TRIAL: NCT00184483
Title: Randomized Multi Site Trial Comparing Lichtensteins Operation and Prolene Hernia System in Inguinal HErnia Repair.
Brief Title: A Multi-site Trial Comparing Lichtensteins Operation and Prolene Hernia System in Inguinal HErnia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Sorlandet Hospital HF (Other Government); Voss Sykehus (Unknown); Haraldsplass Deaconess Hospital (Other); Sykehuset Ostfold (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Norwegian Hernia Study
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Inguinal Hernia
Keywords: Surgery; Lichtenstein; Prolene Hernia System; Postoperative pain; Recurrence
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lichtenstein's operation (Experimental): Patients with a primary unilateral inguinal hernia are randomized to Lichtenstein's operation to repair their groin hernia
  Interventions: Procedure: Lichtenstein's operation
- Prolene Hernia System (Active Comparator): Patients with a primary unilateral inguinal hernia are randomized to Prolene Hernia System to repair their groin hernia
  Interventions: Procedure: Prolene Hernia System

INTERVENTIONS:
Procedure: Lichtenstein's operation — Lichtenstein's operation to repair primary unilateral inguinal hernia
  Arms: Lichtenstein's operation
Procedure: Prolene Hernia System — Prolene Hernia System to repair primary unilateral inguinal hernia
  Arms: Prolene Hernia System

SUMMARY:
Patients with a primary unilateral inguinal hernia are randomized to Lichtenstein's operation or Prolene Hernia System to repair their groin hernia. Follow up for three years with a total number of 4 clinical examinations. End point is postoperative pain and recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Primary unilateral groin hernia in adult

Exclusion Criteria:

* recurrence warfarin treatment bilateral groin hernia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2001-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
pain postoperative | 3 years

SECONDARY OUTCOMES:
Recurrences after groin hernia repair | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Helge E Myrvold, MD PhD, Study Director — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital, Trondheim, Norway